CLINICAL TRIAL: NCT01834755
Title: Physical and Psychological Evaluation of Patients Reaching End Stage Renal Disease : Effects on the Choice of Renal Replacement Therapy
Brief Title: Physical and Psychological Profiles Associated With Patient's Preference for ESRD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-AOI-03
Record Dates: First submitted 2013-02-13; First posted 2013-04-18 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Other): Evaluation of psychological phenotype with several questionnaire (Big Five, EPADV-16), physical activity with a self-administered questionnaire (Baecke) and several test ( SPPB, Handgrip Strengh test, MicroFET 2 Digital Dynamometer)
  Interventions: Other: Evaluation of psychological phenotype

INTERVENTIONS:
Other: Evaluation of psychological phenotype

SUMMARY:
Highlighting the relationship between psychological and physical profiles and patient's preference to better understand the patient's treatment preference and improve the information provided.

DETAILED DESCRIPTION:
CKD is a Public Health Problem with a prevalence of 10% in general population. For patients reaching The making decision to treat ESRD with renal replacement therapy is a complex process and needs to be shared between patients, family, physician and nephrologist.

Systematic Information delivery about several treatments of ESRD is recommended for patients and his family (Hemodialysis, Peritoneal Dialysis, Kidney Transplantation and Conservative treatment). Some studies on the preference of patients for renal replacement therapy reported a choice for PD about 50% while the registers report a low diffusion of PD (around 10%). Since 2009 we propose a systematic information about the different therapeutic options for ESRD and identified some clinical characteristics associated to patient's preference. However we want to know if psychological or physical phenotype is associated to patient's preference.

The objective of the study is to highlight the relationship between psychological and physical profiles and patient's preference to better understand the patient's treatment preference and improve the information provided.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* CKD with estimated GFR below 20 ml/min/1.73m2 without dialysis treatment
* Patient who accepts information delivery about treatments of ESRF
* Patient who accepted and signed the informed consent
* Subject beneficiary of a social security system

Exclusion Criteria:

* Inability to achieve psychological tests
* Inability to achieve physical tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06-27 (Actual); Study Completion 2013-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison of different psychological and physical characteristics according to patients preference | one day
  The measure is composite:
  criteria evaluated for psychological phenotype are: The score of the Big Five test Scale Assess people's perception of autonomy in various life domains (EPADV-16)
  The criteria evaluated for physical phenotype are:
  * Global physical activity assess with self-administered questionnaire of BAECKE.
  * Evaluation of mobility with Short Physical Performance Battery Score (SPPB)
  * Measure of the maximum isometric strenght of the hand with " Handgrip Strengh test"
  * Assessment of musculoskeletal testing of the leg with MicroFET 2 Digital Dynamometer

SECONDARY OUTCOMES:
Clinical characteristics and laboratory values | one day
  Clinical characteristics (age, sex, way of life, education level, QOL, nephropathy, cardio-vascular comorbidity) and laboratory values (haemoglobin, ferritin, css, creatinine, cystatin C, phosphates, calcium, 25OHD3, PTH and CRP) associated with psychological or physical phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MORANNE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Service de Néphrologie, Nice, France